CLINICAL TRIAL: NCT00502671
Title: An Open Label Study to Evaluate the Safety of Xeloda as Adjuvant Monotherapy in Patients Who Have Undergone Surgery for Colon Cancer, Dukes Stage C.
Brief Title: A Study of Xeloda (Capecitabine) as Adjuvant Monotherapy in Patients With Colon Cancer.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20592
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 1250mg/m2 po bid on days 1-14 of each 3 week cycle

SUMMARY:
This single arm study will evaluate the safety profile of Xeloda as monotherapy for adjuvant treatment of colon cancer. All patients will receive Xeloda 1250mg/m2 p.o. twice daily as intermittent treatment (3 week cycles consisting of 2 weeks of treatment followed by 1 week without treatment). The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* colon cancer (Dukes stage C);
* surgery, with no evidence of remaining tumor;
* ECOG performance status of <=1.

Exclusion Criteria:

* previous therapy for currently treated colon cancer;
* any evidence of metastatic disease;
* history of other malignancy within last 5 years;
* clinically significant cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- Russia (37):
  - Arkhangelsk
  - Astrakhan
  - Barnaul
  - Belgorod
  - Chelyabinsk
  - Irkutsk
  - Izhevsk
  - Kaluga
  - Kazan'
  - Kirov
  - Kostroma
  - Krasnodar
  - Kursk
  - Lipetsk
  - Moscow
  - Nizhny Novgorod
  - Novgorod Veliky
  - Obninsk
  - Orenburg
  - Perm
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Salekhard
  - Samara
  - Sashi
  - Smolensk
  - Stavropol
  - Surgut
  - Tollyatti
  - Tomsk
  - Tver'
  - Tyumen
  - Ufa
  - Volgograd
  - Yekaterinburg
  - Yuzhno-Sakhalinsk

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine: Participants with resected Stage III colon cancer (Dukes C) or high-risk Stage II colon cancer (Dukes B) received capecitabine orally (PO) as 1250 milligrams per meter-squared (mg/m^2) twice daily, once in the morning and once at night, in this non-randomized postmarketing safety study. For those with moderate renal insufficiency at Baseline, the initial dose was reduced to 950 mg/m^2 twice daily. Each 3-week cycle comprised 2 weeks of continuous treatment followed by a 1-week break, and treatment continued for up to 8 cycles (24 weeks) or until relapse, new-onset colon cancer, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Capecitabine
Started | 228
Completed | 151
Not Completed | 77
Not completed — Disease Progression | 13
Not completed — Personal Reasons | 22
Not completed — Lost to Follow-up | 7
Not completed — Protocol Violation | 16
Not completed — Adverse Event | 19

BASELINE CHARACTERISTICS:
Population: Safety Population: All enrolled participants who received a dose of study medication.
Groups:
- Capecitabine: Participants with resected Stage III colon cancer (Dukes C) or high-risk Stage II colon cancer (Dukes B) received capecitabine PO as 1250 mg/m^2 twice daily, once in the morning and once at night, in this non-randomized postmarketing safety study. For those with moderate renal insufficiency at Baseline, the initial dose was reduced to 950 mg/m^2 twice daily. Each 3-week cycle comprised 2 weeks of continuous treatment followed by a 1-week break, and treatment continued for up to 8 cycles (24 weeks) or until relapse, new-onset colon cancer, or unacceptable toxicity.
Arm/Group | Capecitabine
Number analyzed (Participants) | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE), Serious AE, or Death Due to an AE
Description: The postmarketing safety profile of capecitabine was evaluated by collection of AEs, clinical laboratory data, vital signs, and other findings from physical examination. Abnormalities in these findings were captured as AEs, defined as any untoward medical occurrence in a study participant regardless of the suspected cause. Serious AEs were those which, at any dose, met one or more of the following criteria: resulted in fatality, were life-threatening, necessitated new or prolonged existing hospitalization, produced persistent or significant disability, resulted in congenital anomaly or birth defect, were considered medically significant, or required intervention to prevent any of the aforementioned outcomes. Those specific serious AEs which resulted in fatality were also reported separately. The percentage of participants with an AE, serious AE, or AE resulting in death was calculated as [number of participants with event divided by number analyzed] multiplied by 100.
Time Frame: Up to 25 weeks (from Baseline to the end of safety follow-up)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 228
percentage of participants
  Any AE | 56.1
  Serious AE | 6.1
  Death due to an AE | 0.4

2. Secondary Outcome: Percentage of Participants With Early Withdrawal or Discontinuation Due to an AE
Description: The postmarketing safety profile of capecitabine was evaluated by collection of AEs, clinical laboratory data, vital signs, and other findings from physical examination. Abnormalities in these findings were captured as AEs, defined as any untoward medical occurrence in a study participant regardless of the suspected cause. The percentage of participants with early withdrawal or treatment discontinuation due to an AE was calculated as [number of participants with event divided by number analyzed] multiplied by 100.
Time Frame: Up to 25 weeks (from Baseline to the end of safety follow-up)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 228
percentage of participants
  Early withdrawal due to an AE | 8.3
  Discontinuation due to an AE | 10.1

ADVERSE EVENTS:
Time Frame: Up to 25 weeks (from Baseline to the end of safety follow-up)
Arm/Group | Capecitabine
Serious Adverse Events (participants affected / at risk) | 14/228
Other Adverse Events (participants affected / at risk) | 81/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=228)
Myocardial infarction (Cardiac disorders) | 2
Abdominal abscess (Gastrointestinal disorders) | 1
Colon cancer (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Palmar-plantar erythrodysaesthesia syndrome (Nervous system disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=228)
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 12
Palmar-plantar erythrodysaesthesia syndrome (Nervous system disorders) | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.